CLINICAL TRIAL: NCT02519647
Title: Comparison of Intubation Conditions Between the Gliderite and the S-Guide in Patients With Simulated Difficult Airways
Brief Title: Comparison of Intubation Conditions Between the Gliderite and the S-Guide
Acronym: S-Guide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Patrick Schoettker,MD PD, MD, PD, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 267/15
Record Dates: First submitted 2015-07-27; First posted 2015-08-11 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Nasal Obstruction; Lumbar Stenosis, Familial
MeSH Terms: conditions — Nasal Obstruction; Lumbar Stenosis, Familial | interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tracheal intubation with Gliderite (Active Comparator): Gliderite will be used for intubation
  Interventions: Device: Tracheal intubation with Gliderite
- Tracheal intubation with S-Guide (Experimental): S-Guide will be used for intubation
  Interventions: Device: Tracheal intubation with S-guide

INTERVENTIONS:
Device: Tracheal intubation with Gliderite — Tracheal intubation with Gliderite
  Arms: tracheal intubation with Gliderite
Device: Tracheal intubation with S-guide — Tracheal intubation with S-guide
  Arms: Tracheal intubation with S-Guide

SUMMARY:
Intubation with an unchanneled videolaryngoscope mandates the use of a stylet. The Gliderite is a stylet specially designed for videolaryngoscopes. The investigators aim to compare the efficacy of a new designed bougie for intubation in patients with simulated difficult airways.

DETAILED DESCRIPTION:
Intubation with an unchanneled videolaryngoscope mandates the use of a stylet. The Gliderite is a stylet specially designed for videolaryngoscopes. The investigators aim to compare the efficacy of a new designed bougie for intubation in patients with simulated difficult airways.

The primary endpoint will be time necessary for intubation, secondary endpoints will be injuries, ease of use and subjective assessment.

ELIGIBILITY:
Inclusion Criteria:

* Surgery necessitating general anesthesia and orotracheal intubation

Exclusion Criteria:

* History or criteria of difficult intubation
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-05-02 (Actual); Study Completion 2016-06-02 (Actual)

PRIMARY OUTCOMES:
Time necessary to intubate | 50 seconds
  Time needed to pass tracheal tube through vocal cords

SECONDARY OUTCOMES:
Standardized questionnaire assessing injury after intubation | 50 seconds
  Assessment of discomfort after procedure
Standardized questionnaire assessing ease of use of the intubation | 50 seconds
  assessment by doctor of ease of intubation
Subjective ease of use of the intubation assessed by questionnaire | 50 seconds
  assessment by doctor of ease of intubation

CONTACTS AND LOCATIONS:
Overall Officials: patrick Schoettker, MD, PD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Dpt of Anesthesiology, University of Lausanne CHUV, Lausanne, Canton of Vaud, Switzerland